CLINICAL TRIAL: NCT07097350
Title: Study on the Effect of Transparent Cap-Assisted Colonoscopy Combined With Computer-Aided Detection in Improving the Detection Rate of Colorectal Adenomas
Brief Title: Transparent Cap-Assisted Colonoscopy Combined With Computer-Aided Detection in Improving the Detection Rate of Colorectal Adenomas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025K239
Record Dates: First submitted 2025-07-13; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Adenoma
Keywords: transparent cap; computer-aided detection; adenoma detection rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer-aided detection alone (Active Comparator): colonoscopy with computer-aided detection alone
  Interventions: Device: computer-aided detection alone
- transparent cap-assisted colonoscopy combined with computer-aided detection (Experimental): transparent cap-assisted colonoscopy combined with computer-aided detection
  Interventions: Device: transparent cap-assisted colonoscopy combined with computer-aided detection

INTERVENTIONS:
Device: computer-aided detection alone — colonoscopy with computer-aided detection
  Arms: computer-aided detection alone
Device: transparent cap-assisted colonoscopy combined with computer-aided detection — transparent cap-assisted colonoscopy combined with computer-aided detection
  Arms: transparent cap-assisted colonoscopy combined with computer-aided detection

SUMMARY:
A prospective, single-center, single-blind, randomized controlled study to compare the effectiveness of transparent cap-assisted colonoscopy combined with computer-aided detection and computer-aided detection alone in improvement of adenoma detection rate

DETAILED DESCRIPTION:
1. Patients are undergone screening or surveillance colonoscopy at the Endoscopy department of Gastrointestinal endoscopy center of Huadong hospital affiliated to Fudan University.
2. Randomize into 2 interventional groups based on Random function of Statistical Package for the Social Sciences (SPSS) 20.0, including (1) Group 1: computer-aided detection alone and (2) Group 2: transparent cap-assisted computer-aided detection.
3. Collecting variables which consist of primary and secodary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged 45-75 years

Exclusion Criteria:

* Patients scheduled for therapeutic colonoscopy as postoperative surveillance after colorectal surgery, post-polypectomy follow-up, or treatment of histologically confirmed polyps
* Patients with highly suspected or pathologically confirmed colorectal cancer
* Patients presenting with alarm symptoms or signs (hematochezia, melena, unexplained anemia or weight loss, palpable abdominal mass, or a positive digital rectal examination)
* Pregnant or breastfeeding women
* Patients with gastrointestinal obstruction
* Patients with inflammatory bowel disease, familial adenomatous polyposis, or serrated polyposis syndrome
* Patients who have taken anticoagulants (e.g., aspirin, warfarin) within 7 days before colonoscopy or who have coagulation disorders
* Patients currently enrolled in another clinical study or who participated in any clinical trial within the past 60 days
* Insertion failure for any reason (e.g., scope cannot pass an obstruction, patient cannot tolerate the procedure) or colonoscopy not reaching the cecum
* A Boston Bowel Preparation Scale (BBPS) score < 6 at scope insertion (inadequate preparation requiring repeat bowel cleansing)
* Use of non-guideline-recommended bowel preparation agents
* Patients undergoing emergency colonoscopy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate | 2 weeks after the procedure

SECONDARY OUTCOMES:
sessile serrated lesion detection rate | 2 weeks after the procedure
advanced adenoma detection rate | 2 weeks after the procedure
polyp detection rate | 2 weeks after the procedure
Clinically Significant Immediate Post-polypectomy Bleeding（CSIPB）rate | immediately after the procedure
  CSIPB was defined as any bleeding not responding to water jet irrigation or STSC and therefore requiring either coagu lation forceps or mechanical clips to achieve hemostasis
Clinically Significant Delayed Post-polypectomy Bleeding（CSDPB）rate | 2 weeks after the procedure
  CSPEB was defined as any bleeding after completion of the procedure requiring emergency room presentation, hospital isation or re-intervention (endoscopy, angiography, surgery).
perforation rate | immediately after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)